CLINICAL TRIAL: NCT03618251
Title: Evaluation of Infarct Volumetric Software in Strokes of Less Than 24 Hours
Brief Title: Automated Volume Assessment of Acute Stroke
Acronym: AVAAS
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: FCD_2017_20
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Stroke, Software Verification, Diffusion Weighted MRI, Neuroimaging
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ischemic stroke: all patients with a suspicion of ischemic stroke
  Interventions: Diagnostic Test: specific MRI sequences

INTERVENTIONS:
Diagnostic Test: specific MRI sequences — MRI with B 2000 of diffusion weighted imaging and the coefficient of apparent diffusion

SUMMARY:
Stroke is a common disease. It is increasingly managed in non-specialized centers.

The volume of the lesion, evaluated on the diffusion weighted imaging, is a prognostic factor of clinical progression and is useful for the treatment decision.

There is therefore a real interest in having a reliable software able to detect the stroke and evaluate the volume of the cerebral infarction. The aim is to provide rapid information to the interventional neuroradiologist and optimize the care of the patient.

The Alberta Stroke Program Early Computed Tomography Score currently used to predict response to treatment divides the territory of the middle cerebral artery. It has a few limitations, it is unreproducible and concerns only the territory of the middle cerebral artery.

Manual volumetry is a long and also not very reproducible technique. The aim of our study is to evaluate the reproducibility and diagnostic performances of the automated segmentation software based on the diffusion weighted imaging sequence, and to compare it to manual and semi-automatic measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for a recent neurological deficit (less than 24 hours), suspected for a stroke.

Non inclusion criteria :

* Pregnant or breastfeeding women
* Patients with absolute contraindications to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: we will include all adult patient with ischemic stroke which have MRI for stroke diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 406 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
Automated volume assessment of acute stroke | 1 hour
  Our objective is to compare several volumetric techniques (manual, semi-manual, automatic) based on the B 2000 of diffusion weighted imaging and the coefficient of apparent diffusion.
  We will also evaluate the correlation between the volumes obtained by the different techniques and the final volume of FLAIR infarction and diffusion in a subgroup of patients for whom a follow-up MRI is feasible.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation A De Rothschild, Paris, France